CLINICAL TRIAL: NCT00003159
Title: Randomized Trial of Surgical Resection With or Without Pre-Operative Chemotherapy in Patients With Operable Non-Small Cell Lung Cancer (NSCLC) of Any Stage
Brief Title: Surgery With or Without Preoperative Chemotherapy in Treating Patients With Resectable Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065952; MRC-LU22; EORTC-08012; EU-97016; ISRCTN25582437
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2005-05

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage 0 non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Cisplatin; Docetaxel; Gemcitabine; Ifosfamide; Mitomycin; Paclitaxel; Vinblastine; Vinorelbine; Neoadjuvant Therapy

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: docetaxel
Drug: gemcitabine hydrochloride
Drug: ifosfamide
Drug: mitomycin C
Drug: paclitaxel
Drug: vinblastine sulfate
Drug: vinorelbine tartrate
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known if surgery is more effective with or without preoperative chemotherapy in treating non-small cell lung cancer.

PURPOSE: This randomized phase III trial is studying surgery and preoperative chemotherapy to see how well they work compared to surgery alone in treating patients with resectable non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the survival of patients with resectable non-small cell lung cancer treated with surgery with or without preoperative chemotherapy.

Secondary

* Compare the quality of life of patients treated with these regimens.
* Compare pre-randomization clinical and post-surgical pathological staging in patients treated with these regimens.
* Compare resectability rates in patients treated with these regimens.
* Compare time to and site of relapse in patients treated with these regimens.
* Determine response in patients treated with preoperative chemotherapy.
* Determine the adverse effects of preoperative chemotherapy in these patients.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo surgical resection no more than 4 weeks after randomization.
* Arm II: Patients receive one of the following chemotherapy regimens immediately after randomization:

  * Regimen 1: Patients receive mitomycin IV, vinblastine IV, and cisplatin IV on day 1.
  * Regimen 2: Patients receive mitomycin IV, ifosfamide IV over 3 hours, and cisplatin IV over 1 hour on day 1.
  * Regimen 3: Patients receive cisplatin IV over 2 hours on day 1 and vinorelbine IV over 5 -10 minutes on days 1 and 8.
  * Regimen 4: Patients receive paclitaxel IV and carboplatin IV on day 1.
  * Regimen 5: Patients receive gemcitabine IV on days 1 and 8 and cisplatin IV over 2 hours on day 1.
  * Regimen 6: Patients receive docetaxel IV and carboplatin IV on day 1. In all regimens, treatment repeats every 3 weeks for a total of 3 courses. Patients undergo surgical resection at least 4 weeks after the last course of chemotherapy.

Quality of life is assessed at 6 and 12 months and then annually thereafter.

Patients are followed 1 month after surgery, 6 months after randomization, every 3 months for 2 years, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 600 patients (300 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven non-small cell lung cancer

  * Resectable disease
  * Previously untreated disease
* No evidence of distant metastases

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 3,000/mm^3
* Neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Considered fit for chemotherapy and surgical resection
* No other disease or prior malignancy that would preclude study treatment
* No active infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent prophylactic colony-stimulating factors (except for secondary prophylaxis)
* No concurrent immunotherapy

Chemotherapy:

* Not specified

Endocrine therapy:

* No concurrent hormonal agents, except corticosteroids

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No other concurrent anticancer therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 1997-08; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Survival

SECONDARY OUTCOMES:
Quality of life as measured by SF-36 questionnaire at baseline, 6 months, 12 months, and then annually thereafter
Clinical and post-surgery pathological staging at pre-randomization
Resectability rates
Extent of surgery
Time to and site of relapse
Tumor response to chemotherapy
Adverse effects of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Hodson — Medical Research Council; Ian E. Smith, MD — Royal Marsden NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Medical Research Council Clinical Trials Unit, London, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England

REFERENCES:
- [Result] Gilligan D, Nicolson M, Smith I, Groen H, Dalesio O, Goldstraw P, Hatton M, Hopwood P, Manegold C, Schramel F, Smit H, van Meerbeeck J, Nankivell M, Parmar M, Pugh C, Stephens R. Preoperative chemotherapy in patients with resectable non-small cell lung cancer: results of the MRC LU22/NVALT 2/EORTC 08012 multicentre randomised trial and update of systematic review. Lancet. 2007 Jun 9;369(9577):1929-37. doi: 10.1016/S0140-6736(07)60714-4. PMID 17544497
- [Result] Hopwood P, Nankivell M, Pugh C, et al.: Impact of pre-operative chemotherapy on the quality of life (QL) of patients with resectable non-small cell lung cancer (NSCLC): experience from the MRC LU22/NVALT/EORTC 08012 multicentre randomised trial. [Abstract] J Clin Oncol 25 (Suppl 18): A-9020, 498s, 2007.
- [Result] Nicolson M, Gilligan D, Smith I, et al.: Pre-operative chemotherapy in patients with resectable non-small cell lung cancer (NSCLC): first results of the MRC LU22/NVALT/EORTC 08012 multi-centre randomised trial. [Abstract] J Clin Oncol 25 (Suppl 18): A-7518, 389s, 2007.